CLINICAL TRIAL: NCT02924714
Title: Discontinuation of Imatinib in Patients With Oligo-metastatic Gastrointestinal Stromal Tumor That Has Become Radiologically Undetectable With Treatment
Brief Title: SSG XXV: The Stop-GIST Trial; Discontinuation of Imatinib in Patients With Oligo-metastatic GIST
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Øyvind Sverre Bruland, Professor in clinical oncology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SSG XXV: Stop-GIST
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Discontinuation of imatinib (Other): Patients treated with imatinib longer than 5 years for oligo-metastatic GIST (≤ 3 metastases) and who have no longer detectable GIST lesions on CT/MRI imaging following complete surgical resection (R0/R1-resection) or RFA of the metastases are assigned to discontinue imatinib.
  Interventions: Other: Discontinuation of imatinib

INTERVENTIONS:
Other: Discontinuation of imatinib

SUMMARY:
The trial "The stop-GIST trial" is an Oslo University Hospital sponsored, prospective, open-label, 1-group, multicenter phase II trial evaluating discontinuation of imatinib in highly selected patients treated with imatinib longer than 5 years for oligo-metastatic GIST (≤ 3 metastases) and who have no detectable overt GIST lesions on CT/MRI imaging following complete surgical resection (R0/R1-resection) or radiofrequency ablation (RFA) of the metastases.

DETAILED DESCRIPTION:
Patients with metastatic GIST are currently recommended to have life-long treatment with tyrosine kinase inhibitors (TKI). The standard first-line treatment is imatinib, which is switched to other drugs at progression or if the patient does not tolerate imatinib. The prevailing hypothesis is that imatinib and other TKIs fail to completely eradicate metastatic GIST and that progression is inevitable if imatinib treatment is discontinued. However, the SSGXVIII/AIO trial found that 3 years of adjuvant imatinib yielded both superior RFS and OS rates compared to 1 year of adjuvant imatinib, which finding does not exclude the hypothesis that sufficiently long administration of imatinib might sometimes eradicate subclinical GIST. Furthermore, a few retrospective studies have reported favorable survival outcomes with surgery of residual disease in metastatic GIST in patients responding to imatinib, and a subset (approximately 20%) of patients with advanced GIST do not progress within the first 10 years on imatinib. Imatinib treatment comes with potential side-effects and, as of now, considerable costs to the society. Therefore, discontinuation of imatinib in highly selected patients, i.e. those who have received imatinib for longer than 5 years and who have undergone metastasectomy of all macroscopic oligometastatic disease, needs to be explored as a novel treatment strategy. Discontinuation might lead to detection of durable complete remissions without imatinib or even cure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18.
2. Morphological and immunohistochemical documentation of GIST (immunostaining for KIT/ (CD117) and/or DOG-1 (anoctamin-1)) must be positive on a tumour sample. Patients with demonstrated mutation in KIT or PDGFRA may be entered to the study despite negative immunostaining for KIT and DOG-1 provided that tumour histology is compatible with GIST.
3. Confirmed metastatic disease by radiology, histology, or both in history.
4. >5.0 years of treatment with imatinib for metastatic disease when the breaks in imatinib administration are taken into account.
5. No more than 3 detectable metastases in the liver and/or in the abdomen on imaging of the abdomen and the pelvis or at surgery during the course of the disease.
6. Macroscopically complete resection of all metastases (either R0 or R1 surgery). Patients who have microscopically infiltrated margins (or suspected microscopical infiltration, R1) are eligible to enter the study. Radiofrequency ablation (RFA) of liver metastases in place of surgery is also allowed. Patients whose oligometastatic disease had disappeared completely so that no remaining target lesion for surgery or RFA can be identified (including absence of residual cyst-like lesions) are allowed to enter the study.
7. Eastern Co-operative Oncology Group (ECOG) performance status ≤ 2.
8. Patient has provided a written, voluntary informed consent prior to study entry and any study-specific procedures.

Exclusion Criteria:

1. Patients with metastases outside of the abdomen (e.g. in the bones or lungs).
2. Not willing to donate tumor tissue and/or blood samples for the molecular studies that aim at predicting of GIST recurrence.
3. Presence of a mutation in SDH, or other evidence for SDH deficiency.
4. Presence of neurofibromatosis-1.
5. R2 resection of the primary tumour or metastasis.
6. Patient with inability to grant reliable informed consent.
7. Inability to comply with the scheduled follow-up.
8. Progressive disease during imatinib or other systemic treatments for GIST, before or after surgery/RFA of the metastases.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2017-01; Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 years
  Three-year progression-free survival (PFS) after discontinuation of imatinib.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Overall survival will be measured from the date of discontinuation of imatinib to the date of death resulting from any cause.
Quality of Life (QoL) | 3 years
  EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, MD PhD, Study Director — Comprehensive Cancer Center Helsinki; Øyvind S Bruland, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] Hompland I, Bruland OS. Can Imatinib Be Safely Withdrawn in Patients with Surgically Resected Metastatic GIST? Anticancer Res. 2015 Nov;35(11):5759-65. PMID 26503996